CLINICAL TRIAL: NCT01096121
Title: Interest of Angiotensin-converting Enzyme Inhibitors on Early Sickle Cell Renal Disease in Children. A Randomized, Double-blind Trial Enalapril vs Placebo.
Brief Title: Angiotensin-converting Enzyme Inhibitors and Early Sickle Cell Renal Disease in Children
Acronym: MADREPIEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough inclusions
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P071222; AOM08052 (Other: Assistance Publique - Hôpitaux de Paris)
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-06

CONDITIONS: Sickle Cell Disease
Keywords: Angiotensin-converting enzyme inhibitors (ACE); Renal disease; Microalbuminemia
MeSH Terms: conditions — Anemia, Sickle Cell; Kidney Diseases | interventions — Enalapril; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Experimental): Enalapril
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Enalapril — * during 1 month : 0,2 mg/kg/day
  * then during 2 months (if no adverse event): 0,35 mg/kg/day
  * and then during 6 months (if no adverse event): 0,5 mg/kg/day
  Arms: 1
Drug: Placebo — Glucose
  Other Names: Glucose
  Arms: 2

SUMMARY:
Patients with sickle cell anaemia may develop renal disease. In fact, renal disease occurred in 40% of adults patients (macroalbuminuria) with evolution to end-stage renal disease for half of them. Microalbuminuria is an early and sensitive marker of glomerular damage. It appears during the first decade and occurred in 20 to 25% of infants (2 to 18 years). Physiopathology of renal scarring is not well understood actually. Renal scarring might be due to glomerular hyperfiltration and vascular and endothelial damage. Angiotensin-converting enzyme inhibitors (ACE) were studied and used in diabetic nephropathy. In a study on 26 sickle cell adults, albuminuria was reduced about 50% by ACE compared to placebo after six months treatment. It might be interesting studying ACE efficacy in sickle cell children with microalbuminuria because renal disease is directly related to sickle cell and is not influenced by other cardiovascular risk factors like in adult patients.

We hypothesized to have a successful ACE treatment in more than 40% of cases after a nine months treatment period. A success is defined as a 50% reduction of the albuminuria/creatinuria ratio.

DETAILED DESCRIPTION:
This is a multicenter study. In order to include 72 patients we should pre-include 400 patients.

They will be included in the study after signing the protocol consent. For final inclusion in the study, two albuminuria/creatinuria ratio should be over or equal to 3mg/mmol. If so, inclusion will be done and patient will be randomized (placebo/enalapril) by CLEANWEB software. A blood sample will be done.

Treatment tolerance will be check up at day 7 (blood sample for renal tolerance and clinical examination), month 1(clinical examination), month 3(clinical examination), month 6(clinical examination), and month 9 (clinical examination). Treatment efficacy will be evaluated by albuminuria/creatinuria ratio at month 1, month 3, month 6, and month 9. Physiopathology of ACE efficacy will be studied at first day and month 9 by dosage of ICAM-1 and VCAM-1.

Treatment plain posology (0.5mg/kg/day) will be progressively obtained on a three months period, beginning at 0.2mg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease (SS, SC, Sb thalassemia, SD Punjab)
* Affiliation to French Health benefits
* Signed informed consent
* Albuminemia / Creatinemia >= 3 mg / mmol (on 2 samples)

Exclusion Criteria:

* Albuminemia / Creatinemia > 100 mg / mmol
* Hypersensibility to enalapril
* Angio-oedemas due to a previous treatment by ACE
* idiopathic or hereditary angio-oedemas
* cerebral echo-doppler
* treatment by lithium digoxine
* treatment by other ACE
* congenital galactosemia
* Pregnancy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percentage of successful treatment of each arm | at 9 months of treatment
  Successful treatment is defined by a reduction by half of the albuminuria/ creatinuria ratio (mg / mmol).

SECONDARY OUTCOMES:
Measure of albuminuria/ creatinuria ratio | at 1, 3 and 6 month of treatment.
Dosage of circulating forms of cell adhesion molecules ICAM-1 and VCAM-1 | at the first day and at 9 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tim ULINSKI, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Trousseau Hospital, Nephro-pediatric unit, Paris, France

REFERENCES:
- [Derived] Sasongko TH, Nagalla S. Angiotensin-converting enzyme (ACE) inhibitors for proteinuria and microalbuminuria in people with sickle cell disease. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD009191. doi: 10.1002/14651858.CD009191.pub4. PMID 34932828